CLINICAL TRIAL: NCT00367900
Title: The Parkinson's, Genes and Environment (PAGE) Study
Brief Title: Parkinson's Genes and Environment Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906093; 06-E-N093
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Parkinson's Disease
Keywords: Diet; Lifestyle; Neurodegenerative Diseases; Elderly Population; Public Health; Parkinson Disease; Environment
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva

GROUPS / COHORTS (1):
- NIH-AARP Diet and Health Study sub study: PAGE: Diet and Health Study members who self-reported a Parkinson's disease (PD) diagnosis on a follow-up questionnaire, and randomly selected controls, will participate in the PAGE sub study.

SUMMARY:
This study will examine the roles of diet, lifestyle, genes, and their possible interactions in the cause of Parkinson's disease, using information from the NIH-AARP Diet and Health Study. The NIH-AARP study was established in 1995 to examine the roles of diet and lifestyle in cancer. It included 567,169 AARP members 50 or older from California, Florida, North Carolina, Pennsylvania, New Jersey, Louisiana, and the Atlanta and Detroit metropolitan areas. In 1995, participants completed a comprehensive questionnaire on diet and a survey on demographics, medications, as well as a follow-up survey in 1996 with more detailed questions on lifestyle and medications, as well as cooking methods and early life dietary habits. A third followup survey is currently underway.

The current NIH-AARP substudy on Parkinson's disease will include approximately 9,000 participants from the NIH-AARP study - 3,000 of whom reported being diagnosed with Parkinson's disease on the most recent survey, and 6,000 control subjects. These study participants provide two saliva samples for genetic analysis and may be asked to complete a telephone interview. In addition, those with Parkinson's disease are asked permission to review medical information regarding their diagnosis.

DETAILED DESCRIPTION:
Parkinson s disease (PD) is the second most prevalent neurodegenerative disease, affecting more than 1 million elderly Americans. The causes of PD are largely unknown, but may include both genetic and environmental factors. We thus propose a large study to investigate the roles of diet, lifestyle, genes and their potential interactions in PD etiology, using the NIH-AARP Diet and Health Study. The AARP cohort was established by investigators at NCI and recruited over half a million participants in 1995 and had prospectively collected detailed information on diet and lifestyle. At baseline, participants were 50 years or older and included 40% women. After more than 8 years of follow-up, we expect to confirm 1,208 incident PD cases with their neurologists. We will comprehensively examine the associations between diet and lifestyle and risk of PD, focusing on dietary antioxidants, fat, caffeine, dairy products, estrogen use, obesity, physical activity, and non steroidal anti-inflammatory drugs (NSAIDs). Further, we will collect saliva samples from PD patients and selected controls without PD for genetic analysis. These results will be used to explore the PD associations with several common genetic polymorphisms and, for the first time, their interactions with several promising diet or lifestyle exposures. Many of the specific aims are novel and important but have been rarely examined in previous investigations. The findings will improve our understanding of the complex relationships among diet, lifestyle, gene-environment interaction, and PD etiology and may potentially contribute to successful PD prevention strategies.

Study Aims:

1. Examine dietary factors that may increase or decrease PD risk.
2. Examine lifestyle factors that may increase or decrease PD risk.
3. Examine genetic polymorphisms in relation to PD risk and their interactions with diet

and lifestyle on PD risk.

Study Population: The NIH-AARP Diet and Health Study cohort.

Design:

1. Longitudinal study for the first two study aims
2. Nested case-control study for the third study aim.

Outcome Parameters: Physician confirmed PD diagnoses.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will be conducted within the infrastructure of the NIH-AARP Diet and Health Study; every participant in the AARP cohort will be eligible for the current investigation. Individuals with PD at baseline (prevalent cases) or with missing information on exposure variables are still eligible for the study, but may be excluded from specific analysis.

The proposed study does not require new recruitment.

EXCLUSION CRITERIA:

No children are included.

The analytic sample includes all participants who respond to the follow-up questionnaires and have non-missing values on the baseline surveys. Participants who reported PD before exposure assessment may be excluded from the analyses.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 3,000 NIH-AARP Diet and Health Study participants who reported a Parkinson's disease (PD) diagnosis on the most recent survey (conducted 2004-2006)and 6,000 control subjects from the cohort who did not report a PD diagnosis.@@@
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2006-08-21 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2014-06-04 (Actual)

PRIMARY OUTCOMES:
Examine factors that increase or decrease risk of PD | duration of study
  Parkinson s disease diagnosis - we validated Parkinson s diagnosis by collecting and reviewing diagnostic information from study participants and their treating physicians. In addition, we collected saliva sample for genetic assays and additional exposure data for analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali Taneja, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Chen H, Zhang SM, Hernan MA, Willett WC, Ascherio A. Diet and Parkinson's disease: a potential role of dairy products in men. Ann Neurol. 2002 Dec;52(6):793-801. doi: 10.1002/ana.10381. PMID 12447934
- [Background] Ascherio A, Zhang SM, Hernan MA, Kawachi I, Colditz GA, Speizer FE, Willett WC. Prospective study of caffeine consumption and risk of Parkinson's disease in men and women. Ann Neurol. 2001 Jul;50(1):56-63. doi: 10.1002/ana.1052. PMID 11456310
- [Background] Chen H, Zhang SM, Hernan MA, Schwarzschild MA, Willett WC, Colditz GA, Speizer FE, Ascherio A. Nonsteroidal anti-inflammatory drugs and the risk of Parkinson disease. Arch Neurol. 2003 Aug;60(8):1059-64. doi: 10.1001/archneur.60.8.1059. PMID 12925360